CLINICAL TRIAL: NCT00074100
Title: Amonafide: Individual Phenotype-Adjusted Chemotherapy for Women With Metastatic Breast Cancer Who Have Progressed Despite Prior Chemotherapy
Brief Title: Amonafide in Treating Women With Metastatic Breast Cancer That Has Progressed After Previous Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: XANTHUS-0001A1-200-GL; MSKCC-03080; CDR0000341687 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-08

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: amonafide dihydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as amonafide, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of amonafide in treating women who have metastatic breast cancer that has progressed after previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the time to progression in women with metastatic breast cancer who have progressed after prior chemotherapy and are now treated with amonafide.
* Determine the overall response rate (complete and partial response) in patients treated with this drug.
* Determine the safety of a phenotypically driven dosing regimen of this drug in these patients.

Secondary

* Determine the time to tumor response, duration of response, and time to treatment failure in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Determine the pharmacokinetic profile of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive amonafide IV over 1 hour on days 1-5. Treatment repeats every 21 days for at least 5 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease may receive additional courses (beyond 5 courses) at the investigator's discretion.

Patients are followed at 30 days and then every 3 months.

PROJECTED ACCRUAL: A total of 175 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic (stage IV) disease
* Relapsed after 1 of the following prior therapy regimens*:

  * Adjuvant therapy containing an anthracycline and a taxane
  * Adjuvant anthracycline therapy followed by first-line metastatic treatment containing a taxane NOTE: *No relapse within 12 months of initiation of prior therapy
* Measurable disease by CT scan or MRI

  * No ascites, pleural effusions, or osteoblastic bone metastases as the only site of measurable disease
* Refractory to hormonal anticancer therapy completed more than 4 weeks before study therapy
* HER2/neu positive allowed provided patient received prior trastuzumab (Herceptin®)

  * MUGA or echocardiogram normal while on trastuzumab
* No known history of or current brain or leptomeningeal metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* No clinically significant abnormal hematological parameters

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN in case of liver metastases)
* AST or ALT no greater than 2.5 times ULN (5 times ULN in case of liver metastases)

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* See Disease Characteristics
* No myocardial infarction within the past 3 months
* No unstable angina pectoris
* No New York Heart Association class III or IV heart disease
* No uncontrolled arrhythmia
* No cardiac insufficiency
* No uncontrolled hypertension
* LVEF at least 50% OR at least lower limit of normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks before, during, and for at least 4 weeks after study participation
* No preexisting neuropathy (motor or sensory) greater than grade 2
* No clinically significant abnormal biochemical parameters
* No clinically significant active infection
* No other prior malignancy except cured nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No other serious illness or medical condition
* No psychological illness or condition that would preclude study participation
* No other known condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* More than 3 months since prior trastuzumab
* More than 2 weeks since prior growth factor therapy (i.e., filgrastim [G-CSF] or sargramostim [GM-CSF])
* No concurrent systemic anticancer immune modulators

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior hormonal therapy
* No concurrent anticancer hormonal therapy
* No concurrent chronic systemic steroids

  * Concurrent topical or inhaled steroids for dermatological or allergy/asthma conditions allowed provided therapy was initiated prior to study enrollment
* Concurrent hormone replacement therapy allowed provided therapy was initiated prior to study enrollment

Radiotherapy

* More than 30 days since prior radiotherapy
* No concurrent radiotherapy directed at target lesions

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* More than 30 days since prior investigational new drug
* More than 2 weeks since prior blood transfusion
* No other concurrent systemic anticancer agents, including immunosuppressive agents
* No other concurrent investigational agents
* Concurrent bisphosphonates allowed provided therapy was initiated prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford A. Hudis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States